CLINICAL TRIAL: NCT04494048
Title: Endoscopic Bariatric Therapies (EBTs): A Retrospective and Prospective Multicenter Registry
Acronym: EBT
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1510016654
Record Dates: First submitted 2020-05-13; First posted 2020-07-31 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Weight Loss; Gastro Esophageal Reflux; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity; Weight Loss; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic Bariatric Therapies (EBT).: patients undergoing Endoscopic Bariatric Therapies
  Interventions: Other: Endoscopic Bariatric Therapies

INTERVENTIONS:
Other: Endoscopic Bariatric Therapies — Participation in this study will allow for data collection through medical chart review for at least 6 standard of care visits up to 1 year after consenting to participate in this registry study. The exposure of interest is total body weight loss, safety and efficacy

SUMMARY:
The purpose of this registry study is to collect data through medical chart review and in patient visits on the efficacy and safety of various Endoscopic Bariatric therapies (EBTs). This is a retrospective and prospective, observational, medical chart review study for at least 6 standard of care visits up to 1 years after a subject consents for study participation.

DETAILED DESCRIPTION:
Endoscopic bariatric therapies such as intragastric balloons, space occupying EBTs, endoscopic sleeve gastroplasty (ESG), primary obesity surgery endolumenal (POSE), and small bowel interventions including gastrointestinal bypass sleeves, etc. are recommended alone or in conjunction with other weight loss treatment modules for patients who cannot or do not want to undergo conventional bariatric surgery or other therapies for obesity (with BMI ≥30 kg/m2) or BMI >27 with comorbidities.

This research is being done in order to find out if endoscopic bariatric therapies work as well as, or better or worse than, other currently available treatment modules to achieve weight loss.

The study is to create a registry to analyze a longitudinal observational cohort of patients who have undergone endobariatric procedures. We will collect information through standard of practice visits and through chart review.

Laboratory data, patient characteristics, imaging, histology will be collected. In certain patients - after specific consent extra blood may be collected for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is considering undergoing EBT for weight loss within 6 months, or has undergone clinically indicated EBT for weight loss within the past 6 months
* Above or equal to 18 years of age.

Exclusion Criteria:

* Any patient who has not undergone or will undergo EBT for weight loss
* Below 18 years of age.

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who will undergo Endoscopic bariatric therapies.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2016-04-05 (Actual); Primary Completion 2035-10-31 (Estimated); Study Completion 2035-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of weight of the various bariatric therapies | Baseline, 1 month, 6 months, and 1 year post procedure
  Compare mean percentage total body weight loss achieved via various Endoscopic Bariatric Therapies compared to baseline, 1 month, 6 months and 1 . year post procedure. This will be calculated by measuring the patients weight on a scale and comparing it to their baseline weight pre procedure.
Safety of procedure measured by in the number of adverse events of procedure | at baseline
  Number of adverse events; Type (unexpected, expected, related, possibly related), frequency and intensity of adverse events at baseline
Safety of procedure measured by in the number of adverse events that occur within 30 days | Within 30 days of the procedure
  Number of adverse events; Type (unexpected, expected, related, possibly related)

SECONDARY OUTCOMES:
Technical success of each bariatric therapy. | through study completion at one year.
  Technical success is the technical success of the procedure.
Change and Improvement in comorbidities | 6 months, 1 year post procedure
  measuring certain anthropometric measurements at baseline and at 6 months and one year. Waist Circumference in cm
Change and Improvement in comorbidities | 6 months, 1 year post procedure
  measuring certain anthropometric measurements at baseline and at 6 months and one year. Blood pressure mmHg
Change and Improvement in comorbidities | 6 months, 1 year post procedure
  measuring certain anthropometric measurements at baseline and at 6 months and one year. These include laboratory measurements (tryglicerides, LDL, A1C, Insulin)
Change in the effect of Endoscopic Bariatric Therapies on reflux | Baseline, 6 months,and 1 year post procedure
  measuring change in gastrointestinal reflux disease (GERD) questionnaire answers
Change in the effect of Endoscopic Bariatric Therapies on reflux | Baseline, 6 months,and 1 year post procedure
  measuring change in ph measurement on ph manometry
Change in the effect of bariatric endoscopic procedure on individuals with fatty liver disease | Baseline, 6 months,and 1 year post procedure
  Measuring change in fibroscan score
Change in the effect of bariatric endoscopic procedure on individuals with fatty liver disease | Baseline, 6 months,and 1 year post procedure
  Measuring change in liver biopsy results
Change in the effect of bariatric endoscopic procedure on individuals with fatty liver disease | Baseline, 6 months,and 1 year post procedure
  Measuring change in liver functions tests (on blood draw alanine alanine aminotransferase (ALT), AST (aspartate aminotransferase) )

CONTACTS AND LOCATIONS:
Overall Officials: Reem Z Sharaiha, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lahooti A, Westerveld D, Johnson K, Aneke-Nash C, Baig MU, Akagbosu C, Hanscom M, Buckholz A, Newberry C, Herr A, Schwartz R, Yeung M, Sampath K, Mahadev S, Kumar S, Carr-Locke D, Aronne L, Shukla A, Sharaiha RZ. Improvement in obesity-related comorbidities 5 years after endoscopic sleeve gastroplasty: a prospective cohort study. Gastrointest Endosc. 2025 Jul;102(1):26-36. doi: 10.1016/j.gie.2024.12.017. Epub 2024 Dec 16. PMID 39694295